CLINICAL TRIAL: NCT06799663
Title: Comparison the Effect of Smart Phones Addiction Between Children and Adolescents on Posture Deviations , Physical Fitness and Intelligence in Egypt
Status: Recruiting | Type: Observational
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Magdy EL-assar, Principal investigator, Kafrelsheikh University
Other Study IDs: KFSIRB200-358
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Smart Phone Addiction
MeSH Terms: interventions — Intelligence Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Comparison the effect of smart phone addiction between children and adolescents on posture , physical fitness and intelligence
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Children
  Interventions: Other: activity questionnaire; Other: Raven's Progressive Matrices test (RPM); Other: Postural assessment software
- Adolescents
  Interventions: Other: activity questionnaire; Other: Raven's Progressive Matrices test (RPM); Other: Postural assessment software

INTERVENTIONS:
Other: activity questionnaire — Physical activity questionnaire will be applied on children and adolescents to compare the effect of smart phone on physical fitness
Other: Raven's Progressive Matrices test (RPM) — Raven's Progressive Matrices test will be applied on children and adolescents to compare the effect of smart phone on intelligence
Other: Postural assessment software — Postural assessment software will be applied on children and adolescents to compare the effect of smart phone on posture

SUMMARY:
Comparison the effect of smart phones addiction between children and Adolescents on posture deviations , physical fitness and intelligence in Egypt

ELIGIBILITY:
Inclusion Criteria:

* Subjects with the following criteria will be enrolled in this study :

The participants will be from middle childhood to adolescents and their age will be ranged from 9to 18 years.

They had Body Mass Index (BMI) = 18.5 :40 . They have a score of 24 or more on the Smart phones addiction scale-short version.

Exclusion Criteria:

* Subjects will be excluded from the study if the participant has the followings that affect that study:

visual or hearing defects, cachexia, any neurological disorders and musculoskeletal problems, any congenital abnormalities .

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents from 9 years to 18 years
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Physical fitness | 2 months
Postural deviation on head and neck | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh university, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared upon the reasonable request from the principal investigator
Supporting Information: Study Protocol, SAP, ICF